CLINICAL TRIAL: NCT04795375
Title: Effects of Physical Activity Counseling After Bariatric Surgery on the Level of Activity and Anthropometric Measures
Brief Title: Physical Activity Counseling After Bariatric Surgery
Status: Unknown | Phase: Not Applicable | Type: Interventional
Last Known Status: Active, not recruiting
Sponsor: Hadassah Medical Organization (Other)
Responsible Party: Principal Investigator, Ram Elazary, Head Bariatric surgeon Hadassah Ein Kerem, Hadassah Medical Organization
Allocation: Randomized | Model: Parallel | Masking: None | Purpose: Supportive Care
Other Study IDs: BPA-0965-HMO
Record Dates: First submitted 2021-03-04; First posted 2021-03-12 (Actual); Last update posted 2022-05-17 (Actual); Status verified 2022-05

CONDITIONS: Obese; Quality of Life; Exercise; Behavior, Health; Bariatric Surgery
Keywords: Physical Activity; Exercise
MeSH Terms: conditions — Obesity; Motor Activity; Health Behavior

STUDY DESIGN:
Oversight: FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- Intervention (Experimental): The intervention group will receive Physical activity counseling and guidance by a certified Nurse during the six months after the surgery, additional to the routine follow-up after bariatric surgery at Hadassah-Ein Kerem Hospital.
  Interventions: Behavioral: Physical Activity counseling
- Control (No Intervention): The control group will receive the routine follow-up followed at Hadassah-Ein Kerem Hospital after bariatric surgery, which includes long term follow-up with the surgeon and a dietitian.
  Participants at the Control group will receive Physical activity counseling by a certified nurse at the end of trial.

INTERVENTIONS:
Behavioral: Physical Activity counseling — The Physical activity counseling techniques will be based on the Self Determination Theory and Five A's (Assess, Advise, Agree, Assist, Arrange). Guidelines for physical activity will include combined aerobic and resistance exercises.
  Each participant in the intervention group will receive personal exercise prescriptions in accordance the post-surgical statues and exercise recommendations after bariatric surgery. Participants will receive long term follow-up and accompaniment during the first six months after the surgery, through Personal meetings with a certified nurse, Phone-calls, motivational massages, and Exercise Videos.
  Arms: Intervention

SUMMARY:
This study will examine whether providing physical activity counseling and guidance to patients post bariatric surgery, along with long-term personal follow-up for six months after the surgery, may increase the level of physical activity, and it's effect on anthropometric and functional measures.

DETAILED DESCRIPTION:
Bariatric surgery is considered to be most effective in treating morbid obesity for patients with BMI≥40 or BMI≥35 with comorbidity for obesity.

postoperative weight loss following any type of bariatric surgery is largely dependent on the extent to which patients can make and sustain changes in their eating habits and activity level. Adopting physical activity habits can help to optimize outcomes after bariatric surgery, such as contributing to the rate of weight loss after the surgery and maintain lean body mass.

In order to successfully implement a behavioral change regarding the adaptation of healthy lifestyle habits in obese patients, it is vital to promote physical activity counseling after the surgery, and to find an effective intervention that can support habitual physical activity.

The aim of this trial is to examine the effect physical activity counseling after bariatric surgery on the amount and intensity of activity performed, quality of life, anthropometric and functional measures during the first year after surgery.

Up to eighty Participants will be recruited for the trial, and will be randomly assigned to one of the two study arms (Control, Intervention). The intervention group will receive physical activity counseling and guidelines for the following six months after the surgery.

All participants will receive a pedometer to track daily steps for 7 days at different time points before and after the intervention. Additional Measurements will be taken at a pre-surgical baseline assessment and throughout the trial, and will include anthropometric measures (Weight, BMI, and body composition) and functional measures (Handgrip, 6-minute walk test, chair stand-up test).

All participants will fill out a the 7-day international Physical Activity questionnaire, Self-efficacy for physical exercise scale, and SF-36 questionnaire, before and after the intervention.

ELIGIBILITY:
Inclusion Criteria:

* BMI ≥ 40 kg/m2 or 35 kg/m2 with comorbidities
* 18 to 50 Years old
* Patient is suitable according to the pre-operative evaluation standards to undergo Bariatric surgery
* Speaks Hebrew/Arabic fluently

Exclusion Criteria:

* Cognitive decline or severe psychiatric or mental illness
* Patient undergone bariatric surgery in the past
* Pregnancy or Breastfeeding
* Orthopedic disease that limits training and mobility (such as severe arthritis, injury or fractures)
* Heart disease with a risk to exercise (heart failure, severe aortic stenosis, uncontrolled arrhythmia, and acute coronary syndrome)
* Moderate /severe lung disease or COPD with FEV1 / FVC <70% on a pulmonary function test

Ages: 18 Years to 50 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult
Enrollment: 49 (Actual)
Dates: Start 2021-03-01 (Actual); Primary Completion 2022-12-30 (Estimated); Study Completion 2023-03-01 (Estimated)

PRIMARY OUTCOMES:
Average daily Step count | change from Baseline at up to 26 weeks (end of the intervention phase)
  Average daily step count of the last 7 days before each visit
Average daily Step count | 1 year post-surgery
  Average daily step count of the last 7 days before each visit
MET's of Self-reported physical activity | Change from Baseline at up to 26 weeks (end of the intervention phase)
  Physical activity score in MET's from self-reported International Physical Activity Questionnaire (IPAQ-sf). Score will be categorized to low, moderate and high intensity level of physical activity.
MET's of Self-reported physical activity | 1 year post-surgery
  Physical activity score in MET's from self-reported International Physical Activity Questionnaire (IPAQ-sf). Score will be categorized to low, moderate and high intensity level of physical activity.

SECONDARY OUTCOMES:
Changes in BMI | Change from Baseline at up to 26 weeks (end of the intervention phase) and 1 year post-surgery
  weight and height will be combined to report BMI in kg/m^2
Changes in Muscle Mass | Change from Baseline at up to 26 weeks (end of the intervention phase) and 1 year post-surgery
  Measuring Muscle mass using bioelectrical impedance analysis scale
six min walk test | Change from Baseline at up to 26 weeks (end of the intervention phase)
  to measure physical funtion,6 min walk test will be assessed in meters
sit to stand test | Change from Baseline at up to 26 weeks (end of the intervention phase) and 1 year post-surgery
  test measuring time of 5 repetitions to assesses functional lower extremity strength
Changes in Handgrip strength test (Kg) | Change from Baseline at up to 26 weeks (end of the intervention phase) and 1 year post-surgery
  to measure the maximum isometric strength of the hand and forearm muscle in KG
changes in Self-efficacy assessed by (SSE)- Self-efficacy for physical exercise scale | Change from Baseline at up to 26 weeks (end of the intervention phase) and 1 year post-surgery
  Self-efficacy score reported in Self-efficacy for physical exercise scale (score 0-90)
Changes in Health-related Quality of life assessed by SF-36 Questionnaire | Change from Baseline at up to 26 weeks (end of the intervention phase)
  reported in Sf-36 Questionnaire
Change in total cholesterol, HDL and LDL levels | Change from Baseline at up to 26 weeks (end of the intervention phase) and 1 year post-surgery
  Results of bloods tests taken at follow-up
Change in glucose and HbA1c levels | Change from Baseline at up to 26 weeks (end of the intervention phase) and 1 year post-surgery
  Results of bloods tests taken at follow-up

CONTACTS AND LOCATIONS:
Locations (1):
- Hadassah Ein Kerem Medical Center, Jerusalem, Israel